CLINICAL TRIAL: NCT02453464
Title: A Phase Ib, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of Humanized Anti-VEGF Monoclonal Antibody(Sevacizumab) Injection Plus FOLFIRI in Chinese Patients With Metastatic Colorectal Cancer
Brief Title: A Phase Ib Study of Humanized Anti-VEGF Monoclonal Antibody (Sevacizumab) Injection Plus FOLFIRI in Chinese Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM129-mCRC-01
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sevacizumab+FOLFIRI (Experimental): Two weeks as one cycle. Cycle 1: FOLFIRI on day1-2, Sevacizumab on day3; Cycle 2 and after: Sevacizumab on day 1, and then FOLFIRI on day1-2
  Interventions: Drug: Sevacizumab; Drug: Irinotecan; Drug: 5-FU; Drug: Leucovorin

INTERVENTIONS:
Drug: Sevacizumab — escalating doses of Sevacizumab : 3mg/kg，4mg/kg，5mg/kg
Drug: Irinotecan — Irinotecan: IV solution, IV over 90 minutes, 180 mg/m², Every 14 days, Until disease progression/toxicity
Drug: 5-FU — 5-FU: IV solution, IV bolus over 2-4 minutes, 400 mg/m²; IV infusion over 46 hours, 2400 mg/m²; Every 14 days, Until disease progression/toxicity
Drug: Leucovorin — Leucovorin: IV solution, IV over 2 hours, 400 mg/m², Every 14 days, Until disease progression/toxicity

SUMMARY:
This is an open-label, multicenter, dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics of Humanized Anti-VEGF Monoclonal Antibody (Sevacizumab) Injection in combination with FOLFIRI in patients with previously treated metastatic colorectal cancer. This study includes two stages. Stage 1 is the dose-escalation stage. Once the maximum tolerated dose (MTD) of Sevacizumab has been established, additional patients will be enrolled in the cohort-expansion stage (Stage 2).

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological confirmed unresectable metastatic colorectal cancer patients who have failed first-line oxaliplatin-based chemotherapy
* At least one measurable lesion (according to RECIST 1.1 )
* At least 4 weeks from the last chemotherapy. If patients received anti-tumor biological products, at least four t1/2 of washout period is needed
* Toxicity from previous treatment has to restore to ≤ grade 1 (NCI CTC4.0)
* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* Adequate hematologic function: ANC ≥ 1.5 × 10^9 /L, HB ≥ 90 g /L (blood transfusion allowed), PLT ≥ 100 ×10^9 /L; Adequate hepatic function: ALT ≤ 2.5 × ULN, AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN (patients with liver metastases ALT ≤ 5 × ULN, AST ≤ 5 × ULN); Adequate renal function: creatinine ≤ 1 × ULN; Coagulation function: INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN
* Patients of childbearing potential (male and female) must agree to use reliable methods of contraception until at least 12 weeks after the last dose
* Patients signed written inform consent
* Willingness and capability to communicate with investigators and to comply with protocol requirements

Exclusion Criteria:

* HCV, TP or HIV antibody positive
* Previously received anti-VEGF protein drugs, such as Bevacizumab,Sevacizumab
* Previously treated with irinotecan
* History of dihydropyrimidine dehydrogenase deficiency
* Patients with alcohol or drug dependence
* Participation in other clinical trials within 4 weeks before enrollment
* Active or chronic hepatitis B infection with HBV DNA > 1.0 * 10^3 IU/mL
* Serious infection requiring intravenous antibiotic therapy
* Symptomatic brain metastases
* Patients with proteinuria at screening (urine protein ≥ 1+)
* History of abdominal fistula, gastrointestinal perforation, abdominal abscess within 6 months prior to enrollment
* History of intestinal obstruction, inflammatory bowel disease, or other intestinal diseases with chronic diarrhea as the major symptom
* Serious non-healing wounds, ulcers or fractures
* Major surgery (excluding biopsy) or significant trauma within 4 weeks prior to enrollment
* Active bleeding within 3 months prior to enrollment
* Bleeding diathesis or coagulation disorder
* History of arterial or venous thrombosis
* History of myocardial infarction or stroke within 6 months prior to enrollment
* Unstable angina, congestive heart failure, New York Heart Association (NYHA) class II heart failure, uncontrollable arrhythmia, uncontrolled hypertension
* Expected to receive surgery during the study or within 1 month after the last dose
* The investigators consider the patients are not suitable for this trial
* Pregnant and lactating women
* Known allergies to any excipient in the study drug
* Patients can not complete this study for any other reason

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 56 days

SECONDARY OUTCOMES:
Adverse Events (NCI-CTC 4.0) | 28 days after the last dose
Plasma pharmacokinetics (PK) parameters for Sevacizumab | Cycle 1(Day3, Day4, Day7, Day10, Day13); Cycle 2-4(Day1);Cycle 4(Day1, Day2, Day5, Day8 ,Day11)
Plasma pharmacokinetics (PK) parameters (Cmax, Tmax, AUC, T1/2) for Irinotecan and its major metabolite SN-38 | Day1, Day2, Day3, Day15, Day16, Day17
Plasma pharmacokinetics (PK) parameters for 5-FU | Day1, Day3, Day15, Day17
Potential biomarkers, including VEGF and ADA | VEGF:Cycle 1(Day3, Day4, Day7, Day10, Day13); Cycle 2-4(Day1);Cycle 4(Day1, Day2, Day5, Day8, Day11); ADA : within 15 minutes before each Sevacizumab administration
Objective Response Rate (ORR) | up to 3 years from date of registration
Disease Control Rate (DCR) | up to 3 years from date of registration
Progression Free Survival (PFS) | up to 3 years from date of registration
Overall Survival (OS) | up to 3 years from date of registration

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The First Hospital of Zhejiang Province, Hangzhou, Zhejiang